CLINICAL TRIAL: NCT01960322
Title: Intervention After MALT (I-AM): Feasibility of Improving Adherence Among Pediatric and Adult Cardiac Transplant Patients Using a Telemetric Intervention
Brief Title: Improving Medication-taking After Liver Transplant
Acronym: I-AM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: University of California, Los Angeles (Other); Children's Hospital Medical Center, Cincinnati (Other); University of Pittsburgh (Other); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 13-0223
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Nonadherence; Tacrolimus; Pediatric Liver Transplant Recipients
Keywords: adherence; nonadherence; compliance; noncompliance; liver transplantation
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Telemetric (Experimental): Enrolled patients will be followed for 12 months during which they will receive the study telemetry intervention.
  Interventions: Behavioral: Telemetric

INTERVENTIONS:
Behavioral: Telemetric — A manualized behavioral management approach focusing on avoidance and addressing barriers to adherence, delivered via telephone or internet chat applications.

SUMMARY:
The specific aim is to pilot-test our developed intervention manual's ability to improve patients' adherence to medications and medical outcomes (rejection rate, liver enzyme levels) in participating centers.

DETAILED DESCRIPTION:
Nonadherence (not taking the medications as prescribed) is the most common cause of late acute rejection in children who have had a liver transplant, and thus is associated with graft loss, increased expenditures on care, and ultimately death. Researchers in this application developed a biomarker to identify nonadherence, calculating the standard deviation (SD) of consecutive immunosuppressant blood levels for each patient to capture the degree of variability between individual levels (higher SD = less consistent levels). By applying a threshold, this marker identifies nonadherent patients. A consortium of transplant centers is currently testing this marker through the MALT (Medication Adherence in children who had a Liver Transplant) study. MALT investigators now propose to take advantage of this existing collaboration to pilot-test an intervention to improve adherence in patients who are identified by this marker.

ELIGIBILITY:
Inclusion Criteria:

* The patient is between 11-19 years of age at enrollment.
* Guardian's consent, child assent (in accordance with each institution's IRB policies).
* The patient is prescribed tacrolimus (either brand or generic formulation).
* The patient has been seen in the enrolling center's clinic at least once in the last two years.
* The patient's SD of tacrolimus was > 2.0 in the year prior to enrollment, with at least 3 levels present to make this determination.
* The patient and at least one guardian speaks English or Spanish at a level that allows her / him to understand the study procedures and consent to the study.

Exclusion Criteria:

* The patient received a liver transplant less than 1 year prior to enrollment.
* The patient has had more than one transplant (including marrow replacement).
* The patient has had biopsy-proven rejection within the past six months.
* The patient has been diagnosed with Hepatitis C.
* The treating physician has instructed the patient not to obtain tacrolimus levels for at least one year in the past year.
* The guardian or child (in a developmentally-appropriate manner) do not understand the study procedures. This will be verified by asking both guardian and child to repeat the study procedures.
* The patient is only seen for consultation - most or all of the child's routine care is provided at another center (or in a community clinic).
* Either the patient or the guardian is actively psychotic or severely disoriented due to any cause, including hepatic encephalopathy (temporary exclusion) or severely mentally retarded as defined in the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV).
* The patient is not medically stable or is hospitalized.

Ages: 11 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2014-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in Adherence | at baseline and one year
  Change in Adherence at one year compared to at baseline measured via the Standard Deviation of Tacrolimus levels obtained

SECONDARY OUTCOMES:
Change in Incidence of rejection | at baseline and at one year
  Change in Incidence of rejection compared at one year to baseline
Liver Enzyme Levels | at baseline
Liver Enzyme Levels | at one year
Feasibility | at one year
  Participation in the intervention (receive all of the remote interactions called for in the manual, presented as a percentage of received / offered during the intervention active phase, 1 year)

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Shemesh, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (3):
  - UCLA Mattell Children's Hospital, Los Angeles, California
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania